CLINICAL TRIAL: NCT07149766
Title: Breast Crawling and Breastfeeding Success
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, öznur tiryaki, Associate Professor, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Zehra Tostanoğlu
Record Dates: First submitted 2025-07-18; First posted 2025-09-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Pregnacy; Newborn; Breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental)
  Interventions: Other: Breast crawling
- Control group (No Intervention)

INTERVENTIONS:
Other: Breast crawling — The newborn will be placed on the mother's abdomen for no more than 60 minutes, during which breast crawling and suckling behaviors will be observed. Throughout this period, the researcher will maintain active communication with the mother, providing information on the importance of breastfeeding.
  The mother will be gently guided to support the baby when necessary, without interfering with the baby's natural instincts. The newborn's heart rate, respiratory rate, and body temperature will be recorded at birth and at the 60th minute.
  Arms: intervention group

SUMMARY:
Breast crawling, also referred to as the newborn's self-attachment, was first observed in 1977 and described as the "first important sucking behavior". During the first hour after birth, the newborn exhibits instinctive movements aimed at locating and attaching to the breast. In 1987, Swedish researchers Widström et al., and later in 1990, Righard and Alade, detailed these behaviors through systematic observation.

They found that when a newborn is placed prone on the mother's abdomen immediately after birth-while the mother is in a supine position-the baby begins to engage rooting and stepping reflexes. These reflexes typically lead the baby to begin crawling toward the breast around 29 minutes after birth, with effective suckling starting approximately 50 minutes postpartum.This instinctual behavior, observed in the first hour of life when the newborn is most alert and active, has been well documented in the literature as "the breast crawl." It demonstrates the neonate's innate capacity to find and latch onto the mother's breast using biological reflexes when uninterrupted.

Righard and Alade emphasized that routine hospital practices often interrupt this natural sequence, which may negatively impact the breastfeeding process. They underlined the importance of preserving the immediate postnatal hour, a critical window in which these behaviors are most likely to occur and support early breastfeeding success.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age,
* Volunteering to participate in the study,
* Ability to speak, write, and understand Turkish,
* No communication difficulties,
* Having had a spontaneous vaginal delivery,
* Primigravida giving birth for the first time,
* The baby was given to the mother within the first hour after birth,
* Having a full-term, singleton, and healthy newborn,
* No condition preventing breastfeeding in either mother or baby.
* The baby was born with an APGAR score of 7 or higher,
* The baby had no tongue, lip, or mouth anomalies,
* Coordination of sucking, rooting, and swallowing was present.

Exclusion Criteria:

* The mother did not want to participate in the study or wished to terminate the study,
* The mother had a postpartum emergency requiring medical intervention.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnacy
Enrollment: 80 (Actual)
Dates: Start 2025-08-25 (Actual); Primary Completion 2025-11-15 (Actual); Study Completion 2025-12-20 (Actual)

PRIMARY OUTCOMES:
Postpartum Comfort Scale | Within the first 24 hours postpartum
  Description: Measures physical, psychological, and environmental comfort after childbirth. (The scale is a 34-item Likert-type scale. The lowest possible score is 34, and the highest is 170. A higher score indicates higher postpartum comfort.)
Postpartum Breastfeeding Self-Efficacy Scale | At 24 hours postpartum
  Description: Evaluates the mother's confidence in her ability to breastfeed successfully. The minimum score that can be obtained from the scale is 14, and the maximum score is 70. The scale has no cut-off point, and a higher score indicates higher breastfeeding self-efficacy.

SECONDARY OUTCOMES:
Demographic Information Form | baseline
  Tool: Mother and Infant Demographic Information Form
  Description: Includes maternal age, parity, delivery mode, gestational week, newborn Apgar scores, birth weight, and gender.
  Purpose: To identify potential confounding variables and describe the study population.

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya University, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
For ethical reasons, patient information may be shared upon reasonable request without revealing their identities for security reasons.